CLINICAL TRIAL: NCT06930872
Title: A Phase 1, Open Label, Drug Interaction Study to Evaluate the Effect of ZYN002 on the Pharmacokinetics of CYP3A4, CYP2C19, CYP2C9, CYP2D6, CYP1A2, CYP2C8, and CYP2B6 Probe Substrates, and Valproate in Healthy Adult Participants
Brief Title: Drug Interaction Study of ZYN002 Transdermal Gel and Probe Substrates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harmony Biosciences Management, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ZYN2-CL-007
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Drug Interaction

STUDY DESIGN:
Intervention Model Description: Part 1: Participants will receive probe substrates in Periods 1 and 3 and ZYN002 treatment in Periods 2 and 3.
  Part 2: Participants will receive probe substrate in Periods 1 and 3 and ZYN002 treatment in Periods 2 and 3.
Masking Description: This is an open-label, 2-part, fixed-sequence DDI study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Interaction of ZYN002 and substrates (Experimental): Substrates: midazolam, omeprazole, losartan, dextromethorphan, caffeine, repaglinide, and bupropion
  Interventions: Drug: Part 1
- Part 2: Interaction of ZYN002 and VPA (Experimental)
  Interventions: Drug: Part 2

INTERVENTIONS:
Drug: Part 1 — ZYN002 (transdermal), midazolam (oral), omeprazole (oral), losartan (oral), dextromethorphan (oral), caffeine (oral), repaglinide (oral), bupropion (oral)
  Other Names: Synthetic cannabidiol (sCBD)
  Arms: Part 1: Interaction of ZYN002 and substrates
Drug: Part 2 — ZYN002 (transdermal), VPA (oral)
  Other Names: sCBD
  Arms: Part 2: Interaction of ZYN002 and VPA

SUMMARY:
This study is an open-label drug-drug interaction (DDI) study of ZYN002 transdermal gel and multiple drugs.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, 2-part, fixed-sequence, 3-period DDI study to evaluate the effect of ZYN002 transdermal gel on the pharmacokinetics (PK) of probe substrates and their metabolites. In addition, this study is designed to evaluate the safety and tolerability of ZYN002 transdermal gel after multiple-dose topical application to healthy adult participants.

Part 1 - DDI with probe substrates for cytochrome P450 (CYP)3A4, CYP2C19, CYP2C9, CYP2D6, CYP1A2 administered as single oral doses followed by the staggered dosing of probe substrates for CYP2C8 and for CYP2B6 administered as single oral doses.

Part 2 - DDI with valproate (valproic acid [VPA]), a probe substrate for β-oxidation and glucuronidation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults, 18-55 years of age, inclusive, at the time of Screening.
2. Judged by the Investigator to be in generally good health at Screening based upon the results of a medical history, physical examination, 12-lead ECG, and clinical laboratory test results. Laboratory results outside of the reference range, but acceptable, must be documented as not clinically significant (NCS) at the discretion of the Investigator.
3. Participants must have a body mass index between 18 and 30 kg/m² at the time of Screening.
4. Females of childbearing potential must have a negative pregnancy test result at the Screening Visit and on Day -1 before admission to the CRU. Females who are not of childbearing potential are defined as being postmenopausal for >=12 months or having a history of hysterectomy and/or bilateral oophorectomy and/or bilateral tubal ligation.

Exclusion Criteria:

1. A) Females who are pregnant, nursing or planning to become pregnant or females of childbearing potential, who are unwilling to use medically acceptable method of contraception or B) Males with a female partner who is pregnant, nursing, or planning to become pregnant or a female partner of childbearing potential who is unwilling to use a medically acceptable method of contraception.
2. Are homozygous for CYP2C19*2 or heterozygous carriers of CYP2C19*2/CYP2C19*3 or CYP2C9*2/CYP2C9*3 or CYP2D6*2/CYP2D6*3 haplotypes categorized as poor metabolizers.
3. Has consumed alcohol 48 hours prior to Day 1 or during the study.
4. Has eaten any food or drink/beverage containing, grapefruit or grapefruit juice, apple, cranberry, Seville orange or orange juice, vegetables from the mustard family (e.g., kale, spinach, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, parsley, mustard greens, endive, red cabbage, asparagus, or mustard), and chargrilled meats within one week prior to study start (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Maximum measure plasma concentration (Cmax) of probe substrates and metabolites | Days 1-3 (Period 1), Days 24-26 (Period 3)
  Blood samples collected at pre dose, and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours post dose.
Cmax of repaglinide and metabolite | Days 3 and 4 (Period 1), Days 26 and 27 (Period 3)
  Blood samples collected at pre dose, and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, and 24 hours post dose.
Cmax of bupropion and metabolite | Days 4-10 (Period 1), Days 27-33 (Period 3)
  Blood samples collected at pre dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 48, 72, 96, 120, and 144 hours post dose.
Cmax of CBD, delta-9-tetrahydrocannabinol (THC), and CBD metabolites | Days 24-33 (Period 3)
  Blood samples collected at pre dose and at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, and 144 hours post dose.
Amount excreted in urine over the collection period (Ae0-12) of CBD and its metabolites | Day 17 (Period 2), Days 24 and 32 (Period 3)
  Urine samples collected over a 12-hour period.
Cmax of VPA and metabolite | Days 1-4 (Period 1), Days 18-21 (Period 3)
  Blood samples collected at pre dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose.
Cmax of CBD, THC, and CBD metabolites | Days 18-21 (Period 3)
  Blood samples collected at pre dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours post dose.
Ae0-12 of VPA and metabolites | Days 1-4 (Period 1), Day 17 (Period 2), Days 18-20 (Period 3)
  Urine samples collected over a 12-hour period.
Ae0-12 of ZYN002 and metabolites | Day 17 (Period 2), Days 18 and 20 (Period 3)
  Urine samples collected over a 12-hour period.

SECONDARY OUTCOMES:
Number of participants with skin irritation in ZYN002 application areas | Up to 33 days
  Skin assessment examination
Number of participants with abnormal physical examination results | Up to 33 days
  Targeted physical examination
Number of participants with abnormal clinical laboratory results | Up to 33 days
  Laboratory testing
Number of participants with abnormal vital sign results | Up to 33 days
  Vital Sign measures
Number of participants with abnormal continuous pulse oximetry results | Up to 33 days
  Continuous pulse oximeter
Number of participants with abnormal electrocardiogram (ECG) | Up to 33 days
  12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polasek, MD, PhD, Principal Investigator — CMAX Clinical Research; Kristen Bzdek, MD, Study Director — Harmony Biosciences Management, Inc.
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia